CLINICAL TRIAL: NCT06532188
Title: Efficacy of Hypno-ear-acupuncture on Insomnia in Advanced Cancer Patients: a Randomized Clinical Trial
Brief Title: Efficacy of Hypno-ear-acupuncture on Insomnia in Advanced Cancer Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 24-001
Record Dates: First submitted 2024-07-29; First posted 2024-08-01 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Oncology; Insomnia; Symptoms and Signs
Keywords: ear acupuncture; medical hypnosis
MeSH Terms: conditions — Neoplasms; Sleep Initiation and Maintenance Disorders; Signs and Symptoms

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Verum (Experimental): Ear acupuncture using permanent needles on predefined acupuncture points followed by a standardized medical hypnosis, needles remain in place for a total of 7 days
  Interventions: Procedure: Hypno-ear-acupuncture
- Sham (Sham Comparator): Ear acupuncture using permanent needles on predefined acupuncture sham points followed by a standardized story without induction of a hypnotic trance, needles remain in place for a total of 7 days
  Interventions: Procedure: Sham Hypno-ear-acupuncture

INTERVENTIONS:
Procedure: Hypno-ear-acupuncture — 5 acupuncture permanent needles on ear acupuncture points according to the National Acupuncture Detoxification Association (NADA) protocol, needle retention after 7 days standardized medical hypnosis:
  * Induction of a trance
  * suggestions for calm and good sleep
  Arms: Verum
Procedure: Sham Hypno-ear-acupuncture — 5 acupuncture permanent needles on ear acupuncture points inserted at non-specific points on the backside of the outer ear, needle retention after 7 days standardized sham hypnosis
  - story without trance induction and suggestions
  Arms: Sham

SUMMARY:
This randomized controlled trial aims to test if a combination of medical hypnosis and ear acupuncture improves sleep quality in patients with advanced cancer during a hospital stay in a palliative care unit.

Patients submitted to our palliative care unit will receive a medical hypnosis and ear acupuncture on the second day of their stay. Sleep quality will be measured using validated patient-reported outcome measures at baseline and after 7 days. Additionally, the use of sleep medication will be documented as a secondary outcome.

The intervention will be compared to a sham medical hypnosis and ear acupuncture to see if the effect of the true intervention has a unique effect.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed cancer
* RCSQ total score <25mm
* ability to read and understand the questionnaires
* ability to give informed consent

Exclusion Criteria:

* pregnancy
* language barrier (non German)
* inability to give informed consent
* hypacusis
* radiographical verified brain metastases
* diagnosed psychosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Richards-Campbell Sleep Questionnaire (RCSQ) | Baseline and after seven days
  Change in Patient-reported outcome measure assessing the sleep quality on five sleep related items using a visual analoge scale Range: 0-100mm (Visual Analog Scale) Domains/items: 5 (Sleep depth, Sleep latency, Awakenings from sleep, Ability to return to sleep, Sleep quality) Total score: mean score of all 5 domains (0-100) Interpretation: higher scores reflect better sleep quality

SECONDARY OUTCOMES:
Edmonton symptom assessment scale (ESAS) | Baseline and after seven days
  Change in Patient-reported outcome measures assessing nine different symptoms on a numerical rating scale Range: 0-10 (Numerical Rating Scale) Domains/items: 9 (pain, fatigue, drowsiness, nausea, annorexia, breathlesness, depression, anxiety, well-being) Total score: mean score of all 9 domains (range: 0-10) Interpretation: higher scores reflect higher symptom burden
Patient health questionnaire 9 (PHQ-9) | Baseline and after seven days
  Change in Patient-reported outcome measure assessing depressive symptoms using 9 items describing the Diagnostic and Statistical Manual of Mental Disorders IV (DSM IV) criteria of depression.
  Range: 0-3 (categorial rating: 0 = "not at all", 3 = "nearly every day" Domains/items: 9 (interest/pleasure in doing things, feeling down or depressed, sleep-related problems, low energy or fatigue, eating problems, self-worth, ability to concentrate, psychomotor problems, thoughts of suicide) Total score: sum of all items (range: 0-27) Interpretation: higher scores reflect higher depressive symptoms
Use of additional medication | From baseline to end of study (total seven days)
  Use of sleep medication (benzodiazepines) and analgesics (opioids, non-opioids, nonsteroidal anti-inflammatory drugs (NSAIDs)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Graz, Graz, Styria, Austria

IPD SHARING:
Plan to Share IPD: No
IPD may be made available on reasonable request

REFERENCES:
- [Background] Ahlberg R, Skarberg K, Brus O, Kjellin L. Auricular acupuncture for substance use: a randomized controlled trial of effects on anxiety, sleep, drug use and use of addiction treatment services. Subst Abuse Treat Prev Policy. 2016 Jul 25;11(1):24. doi: 10.1186/s13011-016-0068-z. PMID 27451854
- [Background] Lam TH, Chung KF, Lee CT, Yeung WF, Yu BY. Hypnotherapy for insomnia: A randomized controlled trial comparing generic and disease-specific suggestions. Complement Ther Med. 2018 Dec;41:231-239. doi: 10.1016/j.ctim.2018.10.008. Epub 2018 Oct 9. PMID 30477846